CLINICAL TRIAL: NCT05293808
Title: Evaluation of Different Doses of Aspirin on Platelet Aggregation in Diabetic Patients With Acute Coronary Syndrome
Brief Title: Platelet Aggregation in Diabetic Patients With Acute Coronary Syndrome Treated With Different Doses of Aspirin
Acronym: DIABE-ASACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giovanni Esposito, Prof., Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8/14
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Acute Coronary Syndrome; Diabetes Mellitus
Keywords: platelet aggregation; acute coronary syndrome; diabetes
MeSH Terms: conditions — Acute Coronary Syndrome; Diabetes Mellitus | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- aspirin 100 mg bis in die (Experimental): aspirin 100 mg twice daily for the first month after acute coronary syndrome
  Interventions: Drug: aspirin 100 mg bis in die
- aspirin 200 mg (Active Comparator): aspirin 200 mg once daily for the first month after acute coronary syndrome
  Interventions: Drug: aspririn 200 mg once daily
- aspririn 100 mg (Active Comparator): aspirin 100 mg once daily
  Interventions: Drug: aspirin 100 mg once daily

INTERVENTIONS:
Drug: aspirin 100 mg bis in die — Patient will be randomized and after 10 days and 30 days we will measure platelets aggregation.
  Arms: aspirin 100 mg bis in die
Drug: aspririn 200 mg once daily — Patient will be randomized and after 10 days and 30 days we will measure platelets aggregation.
  Arms: aspirin 200 mg
Drug: aspirin 100 mg once daily — Patient will be randomized and after 10 days and 30 days we will measure platelets aggregation.
  Arms: aspririn 100 mg

SUMMARY:
Diabetes is an important risk factor of coronary atherosclerosis, and it's well known that platelets of diabetic patients are hyper reactive and so resistant to common antithrombotic therapy. Moreover, in diabetic patients platelets are characterized by high turnover that is responsible of lack of protection by cardioaspirin at common dosage. The aim of our study is to asses the efficacy of different doses of aspirin in diabetic patients with acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with acute coronary syndrome after 24 hours from the coronarography

Exclusion Criteria:

* patients with a family or personal history of bleeding or thrombophilic disorders;
* platelet count >600000/mmc or <150000/mmc
* hematocrit >50% or <25%
* creatinine clearance <30 mL/min

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Effects of different doses of aspirin on platelet aggregation | 1 month
  Valuation of different doses of aspirin once or twice daily on platelet aggregation after 10 day and 30 day from the acute coronary syndrome

SECONDARY OUTCOMES:
Valuation of RAC1 levels in platelets | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Federico II, Naples, Italy